CLINICAL TRIAL: NCT03438292
Title: To Test the Efficacy of Novel Berberine Emulsification by TPGS or Quillaja Extract on the Absorption of Berberine Compared to Berberine Powder in Humans
Brief Title: The Absorption of Bioactive Berberine in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Florida High Tech Corridor Council (Other); Designs for Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB201800017; OCR17000 (Other: University of Florida)
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Berberine; TPGS; Pharmacokinetics; Human intervention study; Quillaja extract
MeSH Terms: interventions — Berberine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A - TPGS emulsified with berberine (Experimental): After an 8-10 hour overnight fast, Group A will receive two soft capsules of TPGS (400mg) emulsified berberine. Following a 7 day wash out period, Group A participants will then receive four capsules of the Quillaja extract emulsified berberine (200mg). Following another 7 day wash out period, Group A participants will then receive two hard shell capsules of the berberine reference powder 400mg. Each TPGS and berberine reference powder capsules contains 400 mg berberine. Each Quillaja extract capsule contains 200 mg berberine. The total amount of berberine throughout is 800 mg.
  Interventions: Dietary Supplement: Berberine; Dietary Supplement: TPGS emulsified berberine; Dietary Supplement: Quillaja extract emulsified berberine
- Group B - Quillaja extract emulsified with Berberine (Experimental): After an 8-10 hour overnight fast, Group B will receive four soft capsules of Quillaja extract emulsified berberine (400mg). Following a 7 day wash out period, Group B participants will then receive two hard shell capsules of the berberine reference powder (400mg). Following another 7 day wash out period, Group B participants will then receive two soft gel capsules of TPGS emulsified berberine (400mg). Each TPGS and berberine reference powder capsules contains 400 mg berberine. Each Quillaja extract capsule contains 200mg berberine. The total amount of berberine throughout is 800 mg.
  Interventions: Dietary Supplement: Berberine; Dietary Supplement: TPGS emulsified berberine; Dietary Supplement: Quillaja extract emulsified berberine
- Group C - Berberine reference powder (Experimental): After an 8-10 hour overnight fast, Group C will receive two hard shell capsules of the berberine reference powder (400mg). Following a 7 day wash out period, Group C participants will then receive two soft gel capsules of TPGS emulsified berberine (400mg). Following another 7 day wash out period, Group C participants will then receive four capsules of the Quillaja extract emulsified berberine (200mg). Each TPGS and berberine reference powder capsules contains 400 mg berberine. Each Quillaja extract capsule contains 200mg berberine. The total amount of berberine throughout is 800 mg.
  Interventions: Dietary Supplement: Berberine; Dietary Supplement: TPGS emulsified berberine; Dietary Supplement: Quillaja extract emulsified berberine

INTERVENTIONS:
Dietary Supplement: Berberine — Two capsules of berberine. Each capsule contains 400 mg berberine. The total amount of berberine throughout is 800 mg.
Dietary Supplement: TPGS emulsified berberine — Two capsules of TPGS/Quillaja extract emulsified berberine. Each capsule contains 400 mg berberine. The total amount of berberine throughout is 800 mg.
  Other Names: Berb-Evail
Dietary Supplement: Quillaja extract emulsified berberine — Four capsules of Quillaja extract emulsified berberine. Each capsule contains 200 mg berberine. The total amount of berberine throughout is 800 mg.

SUMMARY:
Berberine from medicinal plants has therapeutic activities against multiple chronic diseases. But its absorption rate is very low. The objective of this study is to test if adding TPGS or Quillaja extract as an emulsifier enhance the absorption of berberine in human.

DETAILED DESCRIPTION:
Berberine is widely used as an herbal medicine and many health benefits. These well-documented in the literature including lowering blood lipids and glucose, having anti-inflammatory and anti-tumor activity, preventing and delaying neurodegenerative diseases (Alzheimer, Parkinson and Huntington disease) and preventing obesity. However, the absorption rate of berberine is very low. The study team believes adding TPGS or Quillaja extract as an emulsifier enhance the absorption of berberine in human.

The bioavailability of berberine is extremely low. Only 0.5% of orally ingested berberine are absorbed in small intestine and about 0.36% can enter the systemic circulation. About 56% of ingested berberine was not absorbed and additional 43.5% is lost due to metabolism in small intestine.

Vitamin E TPGS (a water-soluble form of vitamin E) is a food additive approved by FDA. It has the potential to increase the absorption of drugs and dietary supplements. TPGS is an effective inhibitor of P-glycoproteins that are responsible for decreased absorption rate of many drugs including berberine. TPGS has the potential be a safe and effective adsorption enhancer for berberine and other bioactive botanicals.

Quillaja extract is a natural GRAS (generally recognized as safe) food-grade surfactant/emulsifier ingredient rich in saponins and sapogenins. It is purified from the Quillaja Saponaria Molina tree which is native to Chile. Quillaja extract is an approved ingredient for use in Food and Beverages by FDA under Title 21 CFR 172.51. It is an approved food additive in the European Union under code E 999. Quillaja extract is an attractive alternative emulsifier for berberine formulation because it meets consumers' demand for natural ingredient. Quillaja extract provides additional benefits of anti-inflammation and cholesterol lowering to dietary supplement. Some early study before 2000 suggested that Quillaja saponin DS-1 promote the absorption of insulin and aminoglycoside antibiotics via the ocular and nasal route by reducing permeability of epithelial barrier. However, it is not known whether quillaja affect absorption of berberine in vivo or in human.

Specific Aims:

1. To determine whether TPGS or Quillaja extract emulsification increase the bioavailability of orally ingested berberine in human volunteers by increasing its plasma concentration time curve (AUC), peak concentration (Cmax), and elimination half time (T1/2).
2. To determine whether TPGS or Quillaja extract emulsification alter phase I metabolism, phase II metabolism, or metabolism by gut microbiota for orally ingested berberine in human

The hypothesis of this research is that TPGS or Quillaja extract emulsification enhances the bioavailability of orally ingested berberine in human by altering it metabolism and pharmacokinetic profiles.

Advertisement will be in the form of flyers. Contact information of investigators will be included in the flyer. All participants will be received written and oral information regarding the natural and potential risks of the study. The informed consent form will be given to the participants to get consent in a private room 7 days before the study.

Screening, Tolerability Test and Informed Consent: Subject will take two capsules of the reference berberine dietary supplement with 8 ounces of room temperature water and subject will remain in a fasted state for 4 hours. After completing 4 hours period, a standard lunch with water will be served. If subject experiences diarrhea after taking supplement, she/he will immediately report to the Principle Investigator, Dr. Wang or the Study coordinator. The result of tolerability test will base on the self-assessment of diarrhea. Twelve participants will be chosen having no symptoms of diarrhea Experiment process: Participants will be advised to avoid berberine, vitamin E TPGS or Quillaja extract supplements and foods, excessive amount of alcohol from the beginning of 7-day run in period to the end of the study.

Participants will receive three treatments (A: TPGS emulsified berberine or B:Quillaja extract emulsified berberine soft gel and C: berberine reference powder in hard shell capsules) using a randomized crossover design. Treatment A, B and C provide an equal amount of berberine at 800 mg dose.

Twelve healthy subjects will be randomly assigned into three groups with 4 in each group. Subjects will be asked to collect initial urine samples in an 8-ounce container provided by the study team before taking the supplement and the rest of urine samples will be collected in a different container after taking supplement for 12 hours period. A trained and certified phlebotomist will be hired to draw blood. A catcher will be implanted in the participants forearm for blood draw. After a baseline blood sample is taken, four participants in group A will receive at two capsules of TPGS emulsified berberine in soft gel (2x400mg) and four subjects in group B will receive four capsules of the Quillaja extract emulsified berberine (4x200mg) in soft shell capsules, and four participants in group C will receive at two capsules of berberine reference powder (2x400mg) in hard shelf. Additional blood samples will be drawn at 0.5 h, 1 h, 2 h, 3h, 4 h, 6 h, 8 h and 12 h for analysis of plasma concentrations of berberine and berberrubine. In addition, the participants will collect all urine samples in a gallon size plastic container during 12 h after the initial dose. A standard breakfast of plain bagel with cream cheese will be given to each participant between 0.5 h and 1 h blood draw. After 4 h blood draw, subjects will be given an identical meal for lunch. Immediately after collection, blood samples will be centrifuged and plasma will be stored at -80 degrees C until analysis. The urine samples will be stored at -80 degrees C until analysis. After two 7-day washout period, the process will be repeated with each group switching over to the other treatment, that is, the group that received treatment A will take treatment B or C and the group that received treatment B will take treatment A or C, the group that received treatment C will take treatment A or B.

Berberine and dihydroberberine in blood exist in nonconjugate free form. A major metabolite berberrubine exists in free form and phase II metabolites including sulfates and glucuronide. In order to analyze berberrubine in all forms, a portion of plasma or urine will be treated with β-glucuronidase from Helix pomatia to hydrolyze its sulfate/glucuronides. Berberine and berberrubine will be extracted from plasma or urine with or without enzyme treatment using solvent or solid phase extraction. The compounds' concentration will be determined using HPLC-ESI-MS/MS method. Pharmacokinetic parameters such as area under the plasma concentration time curve (AUC), peak concentration (Cmax), time at peak concentration (Tmax), and elimination half time (T1/2) will be calculated for berberines, free berberrubine, and total berberrubine. Relative absorption will be expressed as the ratio of calculated AUC's.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal BMI (20-27)

Exclusion Criteria:

* Pregnancy
* Gastro-intestinal conditions
* Diabetics,
* Alcohol and substance abuse history,
* Allergy to berberine,
* Current berberine use,
* Use of H2 blockers, proton pump inhibitors, blood sugar-lowering agents, or statins

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
AUC:the area under the concentration-time curve | Pre-dose, Hour 0.5, Hour 1, Hour 2, Hour 3, Hour 4, Hour 6, Hour 8 and Hour 12
  To determine change in bioavailability of orally ingested berberine in human volunteers by increasing the area under the concentration-time curve (AUC).
Cmax: maximum plasma concentration | Pre-dose, Hour 0.5, Hour 1, Hour 2, Hour 3, Hour 4, Hour 6, Hour 8 and Hour 12
  To determine change in bioavailability of orally ingested berberine in human volunteers by increasing its plasma concentration peak concentration (Cmax).
Tmax: the time point of maximum plasma concentration | Pre-dose, Hour 0.5, Hour 1, Hour 2, Hour 3, Hour 4, Hour 6, Hour 8 and Hour 12
  To determine change in bioavailability of orally ingested berberine in human volunteers by increasing its the time point of maximum plasma concentration (Tmax).

SECONDARY OUTCOMES:
Changes in concentrations of berberine metabolites. | Pre-dose, Hour 0.5, Hour 1, Hour 2, Hour 3, Hour 4, Hour 6, Hour 8 and Hour 12
  To determine change in berberine metabolites concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Gu, PhD, Principal Investigator — Univerisity of Florida; Yavuz Yagiz, PhD, Study Director — Univerisity of Florida; Gary P Wang, MD PhD, FIDSA, Study Director — Univerisity of Florida
Locations (1):
- Food Science and human nutrition department at University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Cai Z, Wang C, Yang W. Role of berberine in Alzheimer's disease. Neuropsychiatr Dis Treat. 2016 Oct 3;12:2509-2520. doi: 10.2147/NDT.S114846. eCollection 2016. PMID 27757035
- [Background] Pirillo A, Catapano AL. Berberine, a plant alkaloid with lipid- and glucose-lowering properties: From in vitro evidence to clinical studies. Atherosclerosis. 2015 Dec;243(2):449-61. doi: 10.1016/j.atherosclerosis.2015.09.032. Epub 2015 Sep 30. PMID 26520899
- [Background] Zou K, Li Z, Zhang Y, Zhang HY, Li B, Zhu WL, Shi JY, Jia Q, Li YM. Advances in the study of berberine and its derivatives: a focus on anti-inflammatory and anti-tumor effects in the digestive system. Acta Pharmacol Sin. 2017 Feb;38(2):157-167. doi: 10.1038/aps.2016.125. Epub 2016 Dec 5. PMID 27917872
- [Background] Wang Y, Shou JW, Li XY, Zhao ZX, Fu J, He CY, Feng R, Ma C, Wen BY, Guo F, Yang XY, Han YX, Wang LL, Tong Q, You XF, Lin Y, Kong WJ, Si SY, Jiang JD. Berberine-induced bioactive metabolites of the gut microbiota improve energy metabolism. Metabolism. 2017 May;70:72-84. doi: 10.1016/j.metabol.2017.02.003. Epub 2017 Feb 10. PMID 28403947
- [Background] Xu JH, Liu XZ, Pan W, Zou DJ. Berberine protects against diet-induced obesity through regulating metabolic endotoxemia and gut hormone levels. Mol Med Rep. 2017 May;15(5):2765-2787. doi: 10.3892/mmr.2017.6321. Epub 2017 Mar 14. PMID 28447763
- [Background] Zou T, Gu L. TPGS emulsified zein nanoparticles enhanced oral bioavailability of daidzin: in vitro characteristics and in vivo performance. Mol Pharm. 2013 May 6;10(5):2062-70. doi: 10.1021/mp400086n. Epub 2013 Apr 26. PMID 23557122
- [Background] Gu S, Cao B, Sun R, Tang Y, Paletta JL, Wu XL, Liu L, Zha W, Zhao C, Li Y, Ridlon JM, Hylemon PB, Zhou H, Aa J, Wang G. Correction: A metabolomic and pharmacokinetic study on the mechanism underlying the lipid-lowering effect of orally administered berberine. Mol Biosyst. 2015 Feb;11(2):664. doi: 10.1039/c4mb90042a. Epub 2014 Dec 23. PMID 25535027